CLINICAL TRIAL: NCT06109415
Title: A Phase 4, Randomized, Blinded, Active-Controlled Study of HTX-011 in Subjects Undergoing Total Shoulder Arthroplasty (TSA)
Brief Title: A Multi-surgery Assessment of ZYNRELEF (HTX-011), AMAZE.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HTX-011-401 (Cohort 1)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain; Total Shoulder Arthroplasty; Multimodal Analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio to HTX-011 or bupivacaine HCl, respectively. All subjects will receive a scheduled postoperative non opioid multimodal analgesic (MMA) regimen.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group 1 Cohort 1 (Experimental): HTX-011 + multimodal analgesic (MMA) regimen
  Interventions: Drug: HTX-011; Drug: Ibuprofen; Drug: Acetaminophen; Device: Luer lock applicator
- Treatment Group 2 Cohort 1 (Active Comparator): Bupivacaine HCl + MMA regimen
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: HTX-011 — 400 mg
  Arms: Treatment Group 1 Cohort 1
Drug: Bupivacaine Hydrochloride — 100 mg
  Arms: Treatment Group 2 Cohort 1
Drug: Ibuprofen — 400 mg
Drug: Acetaminophen — 1 g
Device: Luer lock applicator — Applicator for instillation
  Arms: Treatment Group 1 Cohort 1

SUMMARY:
This is a Phase 4, randomized, blinded, active-controlled, multicohort study to evaluate HTX-011 compared with bupivacaine HCl in subjects undergoing Total Shoulder Arthroplasty (TSA) (Cohort 1).

ELIGIBILITY:
Inclusion Criteria:

* Has American Society of Anesthesiologists (ASA) Physical Status of I, II, or III.
* Is scheduled to undergo a unilateral Total Shoulder Arthroplasty.

Exclusion Criteria:

* Is undergoing a revision surgery.
* Has a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to bupivacaine (or other local anesthetics), NSAIDs, acetaminophen, oxycodone, morphine, or hydromorphone.
* History of severe allergic reaction to aspirin or other NSAIDs, or known history of severe gastrointestinal adverse reactions associated with NSAID use.
* Has taken meloxicam within 10 days prior to the scheduled surgery, or any NSAID within 24 hours prior to the scheduled surgery, with the exception of subjects on low-dose (≤100 mg) daily acetylsalicylic acid for cardioprotection.
* Opioid use for most days within the last 3 months prior to Screening in the opinion of the Investigator.
* Has been administered immediate-release bupivacaine HCl within 5 days prior to the scheduled surgery, or a modified-release bupivacaine product within 14 days prior to the scheduled surgery.
* Has initiated treatment with any of the following medications within 1 month prior to study drug administration: selective serotonin reuptake inhibitors, selective norepinephrine reuptake inhibitors, gabapentin, pregabalin, duloxetine, or cyclooxygenase-2 inhibitors.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to the scheduled surgery (whichever is longer).
* Has a known or suspected history of drug abuse, a positive drug screen (except for cannabinoids) on the day of surgery, or a history of alcohol abuse within the past 5 years.
* Suspected or confirmed active coronavirus disease 2019 (COVID-19) infection.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has undergone 3 or more surgeries within 12 months, other than for diagnostic procedures (eg, colonoscopy).
* Has a body mass index (BMI) >40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Through Day 15

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of bupivacaine and meloxicam | Through 144 hours
Time of occurrence of maximum concentration (Tmax) of bupivacaine and meloxicam | Through 144 hours
Area under the concentration-time curve from Time 0 to the time of the last quantifiable concentration (AUClast) of bupivacaine and meloxicam | Through 144 hours
Area under the concentration-time curve from Time 0 extrapolated to infinity (AUCinf) of bupivacaine and meloxicam | Through 144 hours
Apparent terminal half-life (t½) of bupivacaine and meloxicam | Through 144 hours

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Center for Orthopaedic Reconstruction and Excellence, Jenks, Oklahoma
  - First Surgical Hospital, Bellaire, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - JBR Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided